CLINICAL TRIAL: NCT07219433
Title: Implementing a Mobile Health Application for Women Veterans With Urinary Incontinence: MyHealtheBladder in Function QUERI 3.0 (QUE 25-008)
Brief Title: Implementing a Mobile Health Application for Women Veterans With Urinary Incontinence (MyHealtheBladder): Function QUERI 3.0
Acronym: MHB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 25-003
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Urinary Incontinence
Keywords: Veterans; Implementation Science; Functional Status; Quality of Life; Mobile Applications
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Parallel cluster-randomized trial (parallel-CRT): used in pragmatic evaluations of health program or policy interventions, where half the clusters (in this case, VA sites) are randomly assigned to two interventions: Foundational support only (active comparator) vs. Foundational support plus Reach+Equity Implementation Bundle (experimental).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Foundational Support (Active Comparator): Foundational Support uses the Replicating Effective Program (REP) implementation strategy and includes 5 elements that were developed and tested in our prior Function QUERI work: shareholder engagement, MHB toolkit, Online shared resources (SharePoint) access for clinical program training materials, data reports to assist sites with tracking their data, and Diffusion Networks to promote peer-to-peer sharing and implementation support.
  Interventions: Other: Implementation Strategy: Foundational Support
- Reach+Equity Bundle (Experimental): The Reach+Equity bundle will include the same activities as foundational support plus the Reach+Equity bundle activities which include: 1) external facilitation (provide an outside perspective to help sites identify barriers, develop effective strategies, and navigate complex change processes particularly through the lens of achieving equitable reach); 2) equity in implementation toolkit (guide that supports awareness and consideration of health equity during the implementation process); and 3) equity-focused data-driven monitoring (inform progress regarding equitable reach-related goals).
  Interventions: Other: Implementation Strategy: Reach+Equity Bundle

INTERVENTIONS:
Other: Implementation Strategy: Foundational Support — The primary goal of MHB is to compare implementation approaches while also gathering information on clinical effects of the EBP in its new context. All sites will be randomized to receive 1) foundational REP implementation support alone or 2) foundational REP and Reach+Equity. We propose that low intensity implementation support that promotes engagement with the MHB app (defined as foundational support), will be sufficient for some but not all facilities to successfully incorporate MHB into routine practice.
  Other Names: Foundatiional REP
  Arms: Foundational Support
Other: Implementation Strategy: Reach+Equity Bundle — We hypothesize that adding the Reach+Equity bundle to foundational REP, compared to foundational REP alone, will result in superior implementation outcomes.
  Other Names: Enhanced Support
  Arms: Reach+Equity Bundle

SUMMARY:
Implementing a Mobile Health Application for Women Veterans with Urinary Incontinence (MyHealtheBladder): Function QUERI 3.0 aims to compare implementation approaches while also gathering information on clinical effects of the EBP in its new context and focusing on equitable reach (extent to which the program serves its intended audience). The overall goal is to address a key priority within the implementation science field - identifying and refining metrics for equity and impact. The overall goal is to implement, evaluate, and sustain MyHealtheBladder in 20 VA facilities using a type III effectiveness-implementation hybrid study framework and parallel CRT design.

DETAILED DESCRIPTION:
Background/Purpose. Urinary incontinence (UI) is a highly prevalent condition among women, especially as they age, and can directly impair quality of life, daily function, and long-term independence. Evidence-based behavioral management approaches are first-line treatment for UI; these include treatments such as pelvic floor muscle training, fluid management, and bladder control and voiding strategies. Despite being prevalent and burdensome, UI is often unrecognized and undertreated.

MHB is an interactive mobile health application designed to deliver evidence-based behavioral self-management instruction specifically for women Veterans (WV). In a multi-site RCT (VA IIR HX002827) conducted in VA (n=286) comparing MyHealtheBladder to video visits via VA Video Connect (VVC) delivered by a trained Continence Care provider, MHB resulted in equivalent or greater improvements in UI symptoms and satisfaction compared with VVC. Engagement in MHB was high, with 70% retention and an average of 58 miles saved per Veteran. MHB does not require a clinical visit and has the potential to scale across other VA facilities and generate healthcare savings while maintaining comparable patient-level outcomes to individual clinical encounters.

Objectives. The investigators plan to develop scalable approaches to implement and sustain MyHealtheBladder as well as evaluate reach with foundational support versus the enhanced-implementation strategy (Reach+Equity bundle).

Key questions. How can the Reach+Equity bundle be optimized to implement MHB? What are shareholder perspectives on refinements needed for MHB foundational REP activities, as well as strategies to enhance equitable reach (Reach+Equity bundle)? Are there differences in implementation outcomes (reach, adoption, fidelity, cost) between arms? What are patient-level effectiveness outcomes (urinary symptom severity, quality of life, satisfaction with treatment) among WV who enroll, and do these differ between arms? Are there changes in UI diagnosis rates at implementing sites, and between arms? To address the question: Are there differences in implementation outcomes (reach [primary], fidelity, adoption) between arms? The investigators will use generalized linear models to examine the effect of foundational REP vs. Reach+Equity on implementation outcomes of reach and fidelity at 6, 12, and 18-months (primary). To address the question: Are there differences in effectiveness outcomes (UI severity, QoL, satisfaction) between arms? The investigators will describe effectiveness/quality outcomes for WVs who enroll in MHB, overall and by study arm. Linear mixed effect models including all time points for patient outcomes will be fit to account for clustering of WV within site and repeated measures of patient outcomes.

Methodology. To evaluate implementation, the investigators will randomize sites (n=20) 1:1 to either foundational support or foundational support plus the Reach+Equity bundle. The investigators will use generalized linear models to examine the effect of foundational vs. Reach+Equity on implementation outcomes at 18-months.

ELIGIBILITY:
Inclusion Criteria:

* Women Veterans
* Have any type of Urinary Incontinence existing for at least 3 months

Exclusion Criteria:

* No access to computer or mobile device
* No email account
* Institutionalized

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — MHB is an interactive mobile health application designed to deliver evidence-based behavioral self-management instruction specifically for women Veterans.
Enrollment: 20 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Reach | 18 months
  Reach (primary) will be defined as the percentage of WVs signed up for MHB at the clinic. Although WVs with UI are the target population the investigators do not include the diagnosis in our measure because UI is rarely coded in encounter notes.

SECONDARY OUTCOMES:
Fidelity | 18 months
  Fidelity will be defined as the mean number of sessions completed per enrolled MHB WV.
Adoption | 18 months
  Adoption will be defined as 5 or more enrolled MHB users. The investigators will compute time to adoption for each site.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Goldstein, MD MSPH, Principal Investigator — Durham VA Medical Center, Durham, NC; Alayne D Markland, DO MSc, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be available upon request. Prior to distribution, a local privacy officer and study statistician will certify that the dataset contains no protected health information (PHI). Data will be provided to requestor in electronic format. Sufficient data and descriptors will be made available to duplicate statistical analysis and confirm conclusions in publication. No data or statistical code that could lead to re-identification of individuals will be released. Data will be stored & maintained in an approved, secured location as described in the VA Research Data Inventory Form. The statistician will create de-identified, publication-specific datasets that includes variables from statistical models presented in publication. Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re-identify any individual whose data are included in the dataset.
Supporting Information: Study Protocol
Time Frame: Available upon request.
Access Criteria: Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re- identify any individual whose data are included in the dataset.
URL: https://www.durham.hsrd.research.va.gov/Function_Independence_QUERI.asp